CLINICAL TRIAL: NCT06860113
Title: Evaluation of the T-tilted Position in Retrograde Intrarenal Surgery Using Flexible and Navigable Suction Access Sheath.
Brief Title: Evaluation of Retrograde Intra Renal Surgery in the T-tilted Position
Acronym: RIRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Emad mamdouh adly tawfeik, doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIRS in T-tilted position
Record Dates: First submitted 2025-02-21; First posted 2025-03-05 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Stone, Kidney
Keywords: stone free rate, suction sheath
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard group (Other): Patients will be placed in regular lithotomy position with operating table at 0 degrees of tilting.
  Interventions: Procedure: standard lithotomy position
- T-tilted group (Experimental): Patients will be placed at the T-Tilt position (15 degrees Trendelenburg and 15 degrees away from the surgical side kidney).
  Interventions: Procedure: T-tilting of the patient during surgery

INTERVENTIONS:
Procedure: T-tilting of the patient during surgery — Patients will be placed at the T-Tilt position (15 degrees Trendelenburg and 15 degrees away from the surgical side kidney) during surgery.
  Arms: T-tilted group
Procedure: standard lithotomy position — Patients will be placed in regular lithotomy position with operating table at 0 degrees of tilting.
  Arms: standard group

SUMMARY:
To evaluate the effect of the T-tilted position on the stone-free rate compared to the standard lithotomy position in retrograde intrarenal surgeries.

Common positions include the Trendelenburg position, where the patient is tilted head-down to help gravity move stones from the upper calyces to the renal pelvis, and the modified lateral decubitus position, which improves access to the lower renal poles. A more recent approach, the modified T-tilt position, combines a slight Trendelenburg tilt with lateral positioning, offering optimal access to both the upper and lower calyces while maintaining patient comfort

DETAILED DESCRIPTION:
Retrograde intrarenal surgery is a minimally invasive technique for managing renal stones, especially those in the renal pelvis and calyces. It is the standard of care for renal stones less than 2 cm. Due to the new advancements in endoscopes, ureteral access sheaths, and laser devices,retrograde intra renal surgery has been successful in managing stones with larger sizes.

The stone-free rate following flexible ureteroscopy for renal stones smaller than 2 cm is generally high, with most studies reporting stone free ratio between 80% and 95%.

Variations in stone free ratio can be attributed to factors such as stone composition, location, surgeon experience, intraoperative complications, type of laser and endoscopies Anatomical variations of the kidney especially The stone free ratio is mainly related to stone volume. The more the stone volume and greater risk of residual stones.

suction sheath was developed to enhance the stone free ratio and lower incidence of residual fragments.

Patients position was suggest to lower the postoperative residual rate. Common positions include the Trendelenburg position, where the patient is tilted head-down to help gravity move stones from the upper calyces to the renal pelvis, and the modified lateral decubitus position, which improves access to the lower renal poles. A more recent approach, the modified T-tilt position, combines a slight Trendelenburg tilt with lateral positioning, offering optimal access to both the upper and lower calyces while maintaining patient comfort.

We aimed throughout our study to evaluate the impact of the T-tilted position on stone free rate in retrograde intra renal surgery using flexible suction sheath.

METHODS This study aims to compare two patient positioning techniques during retrograde intrarenal surgery to assess their impact on the stone-free rate. Patients will be randomly assigned to one of two groups: Group A (standard lithotomy position) and Group B (T-Tilt position). The allocation process will use sealed envelopes prepared by an independent third party to ensure unbiased distribution. Both patients and the research team, including data collectors and statisticians, will be blinded to the intervention type to minimize bias. The study will evaluate whether the T-Tilt position improves stone free rate compared to the traditional lithotomy position, potentially optimizing retrograde intra renal surgery outcomes.

Surgical procedure The study will involve a consistent surgical approach to minimize variability. All procedures will be conducted under general anesthesia, with preoperative evaluation based on the American Society of Anesthesiologists physical status classification. Each patient will undergo cystourethroscopy, followed by selective catheterization with a 6F ureteric catheter. The main surgical procedure will be flexible ureteroscopy, performed according to the surgeon's standard technique, without special maneuvers like stone displacement. For patients with large stone burdens, an access sheath will be used to facilitate efficient stone removal. Stone characteristics, including size, location, and renal anatomy, will be recorded for analysis.

At the end of the procedure, an endoscopic examination of the pelvicalyceal system will be performed to assess stone fragmentation and the presence of residual fragments or dust. This examination will be video-recorded for post-operative assessment. The primary outcome of the study will be the comparison of stone free rate between the two positioning groups, while secondary outcomes will include the evaluation of perioperative complications, operative time, postoperative pain, hospital stay, and cost analysis.

ELIGIBILITY:
Inclusion Criteria:

* All patients above the age of 16 years of either sex who did not have a pre-existing ureteral stent presented to the Urology clinic in our university hospitals with kidney stones with size up to 2.5cm (estimated by CTUT as the greatest dimension or the summation of the greatest dimensions).

Exclusion Criteria:

* Previous open renal surgery or renal trauma.
* Patients with renal anomalies.
* Patients with untreated or active UTI.
* Patients who suffer from medical conditions that preclude the application of Trendelenburg position (lung disease, congestive heart failure).

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
stone free rate in the T-tilted position during surgery | the duration of the study of at least 6 months
  Follow up visits will be scheduled after 2 weeks; computed tomography urinary tract (CTUT) will be performed to identify stone-free rates and the procedure will be considered successful if no stones can be identified >4mm.

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams university hospitals, Cairo, Abbassia, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Yuan Y, Liang YN, Li KF, Ho YR, Wu QL, Zhao Z. A meta-analysis: retrograde intrarenal surgery vs. percutaneous nephrolithotomy in children. Front Pediatr. 2023 May 2;11:1086345. doi: 10.3389/fped.2023.1086345. eCollection 2023. PMID 37205217
- [Background] Liaw CW, Khusid JA, Gallante B, Bamberger JN, Atallah WM, Gupta M. The T-Tilt Position: A Novel Modified Patient Position to Improve Stone-Free Rates in Retrograde Intrarenal Surgery. J Urol. 2021 Nov;206(5):1232-1239. doi: 10.1097/JU.0000000000001948. Epub 2021 Jul 12. PMID 34251886
- [Background] Pan J, Xue W, Xia L, Zhong H, Zhu Y, Du Z, Chen Q, Huang Y. Ureteroscopic lithotripsy in Trendelenburg position for proximal ureteral calculi: a prospective, randomized, comparative study. Int Urol Nephrol. 2014 Oct;46(10):1895-901. doi: 10.1007/s11255-014-0732-z. Epub 2014 May 14. PMID 24824146
- [Background] Hyams ES, Munver R, Bird VG, Uberoi J, Shah O. Flexible ureterorenoscopy and holmium laser lithotripsy for the management of renal stone burdens that measure 2 to 3 cm: a multi-institutional experience. J Endourol. 2010 Oct;24(10):1583-8. doi: 10.1089/end.2009.0629. PMID 20629566